CLINICAL TRIAL: NCT01122030
Title: A Randomized, Double-Blind, Placebo-Controlled, Single-Ascending Dose Study to Evaluate the Safety and Efficacy of S-297995 for the Treatment of Opioid-Induced Bowel Dysfunction in Subjects With Chronic Pain
Brief Title: Study to Evaluate the Safety and Efficacy of Naldemedine (S-297995) for the Treatment of Opioid-Induced Bowel Dysfunction in Subjects With Chronic Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 1007V9214
Record Dates: First submitted 2010-05-10; First posted 2010-05-12 (Estimated); Results first posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2011-09

CONDITIONS: Opioid Induced Bowel Dysfunction
Keywords: Chronic pain; Opioid physical dependence
MeSH Terms: conditions — Opioid-Induced Constipation; Chronic Pain | interventions — naldemedine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Cohort 1 (Experimental): In this cohort 9 participants received one 0.1 mg naldemedine tablet and 3 participants received matching placebo administered on Day 15 under fasted conditions.
  Interventions: Drug: Naldemedine; Drug: Placebo
- Cohort 2 (Experimental): In this cohort 9 participants received a single dose of 0.3 mg naldemedine tablets and 3 participants received matching placebo tablets administered on Day 15 under fasted conditions.
  Interventions: Drug: Naldemedine; Drug: Placebo
- Cohort 3 (Experimental): In this cohort 9 participants received a single dose of 1 mg naldemedine tablets and 3 participants received matching placebo tablets administered on Day 15 under fasted conditions.
  Interventions: Drug: Naldemedine; Drug: Placebo
- Cohort 4 (Experimental): In this cohort 9 participants received a single dose of 3 mg naldemedine tablets and 3 participants received matching placebo tablets administered on Day 15 under fasted conditions.
  Interventions: Drug: Naldemedine; Drug: Placebo
- Cohort 5 (Experimental): In this cohort 9 participants received a single dose of 0.03 mg naldemedine oral solution and 3 participants received matching placebo oral solution administered on Day 15 under fasted conditions.
  Interventions: Drug: Naldemedine; Drug: Placebo
- Cohort 6 (Experimental): In this cohort 9 participants received a single dose of 0.01 mg naldemedine oral solution and 3 participants received matching placebo oral solution administered on Day 15 under fasted conditions.
  Interventions: Drug: Naldemedine; Drug: Placebo

INTERVENTIONS:
Drug: Naldemedine — Tablets or solution for oral administration
  Other Names: S-297995; Symproic®
Drug: Placebo — Tablets or solution for oral administration

SUMMARY:
The primary objective of the study is to evaluate the safety of single doses of oral naldemedine in adults physically dependent on opioids.

DETAILED DESCRIPTION:
A single dose of naldemedine or matching placebo will be administered orally to each cohort of 12 participants (9 treatments, 3 placebos) in the morning of Day 15 under fasted conditions. The first cohort will receive a 0.1 mg dose. Cohorts will continue to be enrolled at the next higher dose level until the highest dose level (3 mg) has been achieved or until the study is discontinued due to adverse events or Clinical Opioid Withdrawal Score of >8. A 0.03 mg dose will also be tested. A 0.01 mg dose will be tested if 4 or more subjects experience 1 or more bowel movements within the 24 hour period post dose in the 0.03 mg dosing cohort.

ELIGIBILITY:
Inclusion Criteria:

* Understand and sign an informed consent form
* Males will agree to use an approved double-barrier method of contraception from Day 1 until 1 month after study completion
* Subject tests negative on urine drug test unless the subject has a prescription for the drug(s) that test positive

Exclusion Criteria:

* Subjects under opioid therapy for cancer-related pain or for the management of drug addiction
* Fecal incontinence, irritable bowel syndrome, inflammatory bowel disease, or other active medical disorders associated with diarrhea, intermittent loose stools, or constipation
* Subjects who have participated in any other investigational drug study within 30 days prior to Day 1
* Prior exposure to S-297995

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2010-05-19 (Actual); Primary Completion 2011-02-23 (Actual); Study Completion 2011-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shionogi Clinical Trials Administrator Clinical Support Help Line, Study Director — Shionogi
Locations (1):
- Shionogi Research Site, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at a single study center in the United States.
Pre-assignment Details: Participants were randomized to naldemedine or placebo, screened for 13 days (Days 1-13), and admitted to the clinic on Day 14 for pre-admission assessments. Six cohorts were sequentially enrolled from Cohort 1 (0.1 mg) to Cohort 2 (0.3 mg), Cohort 3 (1 mg), and Cohort 4 (3 mg), and subsequent de-escalation in Cohorts 5 (0.03 mg) and 6 (0.01 mg).
Groups:
- Pooled Placebo: Participants received a single dose of matching placebo administered orally on Day 15 under fasted conditions.
- Naldemedine 0.01 mg: Participants received a single dose of 0.01 mg naldemedine oral solution administered on Day 15 under fasted conditions.
- Naldemedine 0.03 mg: Participants received a single dose of 0.03 mg naldemedine oral solution administered on Day 15 under fasted conditions.
- Naldemedine 0.1 mg: Participants received one 0.1 mg naldemedine tablet administered on Day 15 under fasted conditions.
- Naldemedine 0.3 mg: Participants received a single dose of 0.3 mg naldemedine tablets administered on Day 15 under fasted conditions.
- Naldemedine 1 mg: Participants received a single dose of 1 mg naldemedine tablets administered on Day 15 under fasted conditions.
- Naldemedine 3 mg: Participants received a single dose of 3 mg naldemedine tablets administered on Day 15 under fasted conditions.
Period: Overall Study
Arm/Group | Pooled Placebo | Naldemedine 0.01 mg | Naldemedine 0.03 mg | Naldemedine 0.1 mg | Naldemedine 0.3 mg | Naldemedine 1 mg | Naldemedine 3 mg
Started | 18 | 9 | 9 | 9 | 9 | 9 | 9
Received Treatment | 18 | 9 | 9 | 9 | 9 | 9 | 9
Completed | 18 | 9 | 9 | 9 | 9 | 9 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pooled Placebo | Naldemedine 0.01 mg | Naldemedine 0.03 mg | Naldemedine 0.1 mg | Naldemedine 0.3 mg | Naldemedine 1 mg | Naldemedine 3 mg | Total
Number analyzed (Participants) | 18 | 9 | 9 | 9 | 9 | 9 | 9 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.7 (8.55) | 41.4 (12.99) | 45.2 (13.13) | 45.6 (6.02) | 39.7 (10.64) | 36.6 (10.19) | 44.8 (9.09) | 43.3 (10.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 7 | 5 | 6 | 4 | 2 | 38
  Male | 11 | 2 | 2 | 4 | 3 | 5 | 7 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 5
  Not Hispanic or Latino | 16 | 8 | 8 | 9 | 8 | 9 | 9 | 67
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  White | 18 | 8 | 9 | 9 | 8 | 9 | 9 | 70

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Severity of adverse events (AEs) was graded according to the following definitions:
  * Mild: The subject experiences awareness of symptoms but these are easily tolerated or managed without specific treatment
  * Moderate: The subject experiences discomfort enough to cause interference with usual activity, and/or the condition requires specific treatment
  * Severe: The subject is incapacitated with inability to work or do usual activity, and/or the event requires significant treatment measures.
  The relationship of the event to the study drug was determined by the investigator.
  A serious adverse event (SAE) is defined as any AE occurring at any dose that resulted in any of the following outcomes: death, life-threatening AE, hospitalization or prolongation of existing hospitalization, a persistent or significant disability/incapacity, or a congenital anomaly/birth defect.
Time Frame: From the first dose of study drug on Day 15 up to Day 24.
Population: All participants who received any amount of study drug (safety population).
Measure: Number; unit: participants
Arm/Group | Pooled Placebo | Naldemedine 0.01 mg | Naldemedine 0.03 mg | Naldemedine 0.1 mg | Naldemedine 0.3 mg | Naldemedine 1 mg | Naldemedine 3 mg
Number analyzed (Participants) | 18 | 9 | 9 | 9 | 9 | 9 | 9
participants
  Any adverse event | 9 | 6 | 6 | 5 | 9 | 9 | 9
  Mild adverse events | 9 | 6 | 6 | 4 | 6 | 5 | 1
  Moderate adverse events | 0 | 0 | 0 | 1 | 3 | 3 | 2
  Severe adverse events | 0 | 0 | 0 | 0 | 0 | 1 | 6
  Treatment-related adverse events | 6 | 5 | 3 | 1 | 9 | 8 | 9
  Deaths | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Serious adverse events | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Adverse events leading to discontinuation | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Change From Baseline to 24 Hours Post-dose in Number of Spontaneous Bowel Movements (SBMs) Per Day
Description: Participants completed a bowel function assessment daily diary to record information about bowel movements and constipation. A spontaneous bowel movement was defined as a bowel movement where no laxative or enema was used in the 24 hours preceding the bowel movement.
  Baseline was defined as the average number of SBMs per day during the 2 weeks prior to receiving study drug (Day 1 to Day 15).
Time Frame: Baseline (Day 1 to Day 15) and Day 15 to 16 (0 to 24 hours post-dose)
Population: All randomized participants who received study drug and had at least 1 post-dose efficacy assessment completed (intent-to-treat population). Last observation carried forward (LOCF) imputation was used.
Measure: Mean (Standard Deviation); unit: spontaneous bowel movements / day
Arm/Group | Pooled Placebo | Naldemedine 0.01 mg | Naldemedine 0.03 mg | Naldemedine 0.1 mg | Naldemedine 0.3 mg | Naldemedine 1 mg | Naldemedine 3 mg
Number analyzed (Participants) | 18 | 9 | 9 | 9 | 9 | 9 | 9
spontaneous bowel movements / day
  Baseline | 0.15 (0.13) | 0.20 (0.14) | 0.24 (0.09) | 0.13 (0.13) | 0.17 (0.12) | 0.13 (0.09) | 0.23 (0.11)
  24 hours post-dose | 0.44 (0.51) | 0.11 (0.33) | 0.67 (0.71) | 0.56 (0.73) | 2.00 (1.32) | 3.89 (3.06) | 5.00 (2.12)
  Change from Baseline to 24 hours post-dose | 0.29 (0.48) | -0.09 (0.41) | 0.42 (0.72) | 0.43 (0.68) | 1.83 (1.34) | 3.76 (3.06) | 4.77 (2.15)
Statistical Analysis 1: Comparison: Pooled Placebo vs Naldemedine 0.01 mg; Test type: Superiority or Other; p = 0.0767, ANCOVA; P-values are from a non-parametric rank ANCOVA model with effects for dose group and gender, and baseline number of SBMs as a covariate
Statistical Analysis 2: Comparison: Pooled Placebo vs Naldemedine 0.03 mg; Test type: Superiority or Other; p = 0.8727, ANCOVA; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Pooled Placebo vs Naldemedine 0.1 mg; Test type: Superiority or Other; p = 0.6373, ANCOVA; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Pooled Placebo vs Naldemedine 0.3 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Pooled Placebo vs Naldemedine 1 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: Pooled Placebo vs Naldemedine 3 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 1]

3. Secondary Outcome: Change From Baseline to 48 Hours Post-dose in the Number of SBMs Per Day
Description: Participants completed a bowel function assessment daily diary to record information about bowel movements and constipation. A spontaneous bowel movement was defined as a bowel movement where no laxative or enema was used in the 24 hours preceding the bowel movement. Baseline was defined as the average number of SBMs per day during the 2 weeks prior to receiving study drug (Day 1 to Day 15). Forty-eight hours post-dose was defined as the average number of SBMs per day from 0 to 48 hours post-dose.
Time Frame: Baseline (Day 1 to Day 15) and Day 15 to Day 17 (0 to 48 hours post-dose)
Population: Intent-to-treat population; LOCF imputation was used
Measure: Mean (Standard Deviation); unit: Spontaneous bowel movements / day
Arm/Group | Pooled Placebo | Naldemedine 0.01 mg | Naldemedine 0.03 mg | Naldemedine 0.1 mg | Naldemedine 0.3 mg | Naldemedine 1 mg | Naldemedine 3 mg
Number analyzed (Participants) | 18 | 9 | 9 | 9 | 9 | 9 | 9
Spontaneous bowel movements / day
  Baseline | 0.15 (0.13) | 0.20 (0.14) | 0.24 (0.09) | 0.13 (0.13) | 0.17 (0.12) | 0.13 (0.09) | 0.23 (0.11)
  48 hours post-dose | 0.36 (0.33) | 0.44 (0.39) | 0.67 (0.61) | 0.39 (0.49) | 1.06 (0.68) | 2.28 (1.80) | 2.67 (1.03)
  Change from Baseline to 48 hours post-dose | 0.21 (0.32) | 0.24 (0.39) | 0.42 (0.65) | 0.26 (0.45) | 0.88 (0.68) | 2.15 (1.81) | 2.44 (1.05)
Statistical Analysis 1: Comparison: Pooled Placebo vs Naldemedine 0.01 mg; Test type: Superiority or Other; p = 0.8982, ANCOVA; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Pooled Placebo vs Naldemedine 0.03 mg; Test type: Superiority or Other; p = 0.4946, ANCOVA; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Pooled Placebo vs Naldemedine 0.1 mg; Test type: Superiority or Other; p = 0.9301, ANCOVA; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Pooled Placebo vs Naldemedine 0.3 mg; Test type: Superiority or Other; p = 0.0047, ANCOVA; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Pooled Placebo vs Naldemedine 1 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: Pooled Placebo vs Naldemedine 3 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 1]

4. Secondary Outcome: Change From Baseline to 24 Hours Post-dose in Number of Bowel Movements (BM) Per Day
Description: Participants completed a bowel function assessment daily diary to record information about bowel movements and constipation. Baseline was defined as the average number of BMs per day during the 2 weeks prior to receiving study drug (Day 1 to Day 15).
Time Frame: Baseline and 24 hours post-dose
Population: Intent-to-treat; LOCF imputation was used
Measure: Mean (Standard Deviation); unit: bowel movements / day
Arm/Group | Pooled Placebo | Naldemedine 0.01 mg | Naldemedine 0.03 mg | Naldemedine 0.1 mg | Naldemedine 0.3 mg | Naldemedine 1 mg | Naldemedine 3 mg
Number analyzed (Participants) | 18 | 9 | 9 | 9 | 9 | 9 | 9
bowel movements / day
  Baseline | 0.35 (0.18) | 0.34 (0.10) | 0.41 (0.22) | 0.35 (0.17) | 0.33 (0.12) | 0.29 (0.09) | 0.38 (0.19)
  24 hours post-dose | 0.50 (0.62) | 0.11 (0.33) | 0.67 (0.71) | 0.56 (0.73) | 2.00 (1.32) | 3.89 (3.06) | 5.00 (2.12)
  Change from Baseline to 24 hours post-dose | 0.15 (0.65) | -0.23 (0.36) | 0.25 (0.75) | 0.21 (0.76) | 1.67 (1.35) | 3.60 (3.10) | 4.62 (2.06)
Statistical Analysis 1: Comparison: Pooled Placebo vs Naldemedine 0.01 mg; Test type: Superiority or Other; p = 0.1334, ANCOVA; P-value is from a non-parametric rank ANCOVA model with effects for dose group and gender, and baseline number of BMs as a covariate
Statistical Analysis 2: Comparison: Pooled Placebo vs Naldemedine 0.03 mg; Test type: Superiority or Other; p = 0.3320, ANCOVA; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Pooled Placebo vs Naldemedine 0.1 mg; Test type: Superiority or Other; p = 0.9371, ANCOVA; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: Pooled Placebo vs Naldemedine 0.3 mg; Test type: Superiority or Other; p = 0.0002, ANCOVA; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 5: Comparison: Pooled Placebo vs Naldemedine 1 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 6: Comparison: Pooled Placebo vs Naldemedine 3 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 4, analysis 1]

5. Secondary Outcome: Change From Baseline to 48 Hours Post-dose in Number of Bowel Movements Per Day
Description: Participants completed a bowel function assessment daily diary to record information about bowel movements and constipation. Baseline was defined as the average number of BMs per day during the 2 weeks prior to receiving study drug (Day 1 to Day 15). Forty-eight hours post-dose was defined as the average number of BMs per day from 0 to 48 hours post-dose.
Time Frame: Baseline and 48 hours post-dose
Population: Intent-to-treat population; LOCF imputation was used
Measure: Mean (Standard Deviation); unit: bowel movements / day
Arm/Group | Pooled Placebo | Naldemedine 0.01 mg | Naldemedine 0.03 mg | Naldemedine 0.1 mg | Naldemedine 0.3 mg | Naldemedine 1 mg | Naldemedine 3 mg
Number analyzed (Participants) | 18 | 9 | 9 | 9 | 9 | 9 | 9
bowel movements / day
  Baseline | 0.35 (0.18) | 0.34 (0.10) | 0.41 (0.22) | 0.35 (0.17) | 0.33 (0.12) | 0.29 (0.09) | 0.38 (0.19)
  48 hours post-dose | 0.50 (0.51) | 0.61 (0.49) | 0.72 (0.71) | 0.56 (0.46) | 1.06 (0.68) | 2.28 (1.80) | 2.67 (1.03)
  Change from baseline to 48 hours post-dose | 0.15 (0.53) | 0.27 (0.51) | 0.31 (0.67) | 0.21 (0.52) | 0.72 (0.70) | 1.99 (1.82) | 2.29 (0.98)
Statistical Analysis 1: Comparison: Pooled Placebo vs Naldemedine 0.01 mg; Test type: Superiority or Other; p = 0.7978, ANCOVA; P-values are from a non-parametric rank ANCOVA model with effects for dose group and gender, and baseline number of BMs as a covariate
Statistical Analysis 2: Comparison: Pooled Placebo vs Naldemedine 0.03 mg; Test type: Superiority or Other; p = 0.7143, ANCOVA; [statistical method as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Pooled Placebo vs Naldemedine 0.1 mg; Test type: Superiority or Other; p = 0.7531, ANCOVA; [statistical method as in outcome 5, analysis 1]
Statistical Analysis 4: Comparison: Pooled Placebo vs Naldemedine 0.3 mg; Test type: Superiority or Other; p = 0.0283, ANCOVA; [statistical method as in outcome 5, analysis 1]
Statistical Analysis 5: Comparison: Pooled Placebo vs Naldemedine 1 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 5, analysis 1]
Statistical Analysis 6: Comparison: Pooled Placebo vs Naldemedine 3 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 5, analysis 1]

6. Secondary Outcome: Change From Baseline to 24 Hours Post-dose in Number of Complete Spontaneous Bowel Movements (CSBMs) Per Day
Description: Participants completed a bowel function assessment daily diary to record information about bowel movements and constipation. A complete spontaneous bowel movement was defined as a bowel movement where no laxative or enema was used and the bowel movement resulted in a sensation of complete evacuation (based on the question of "having a feeling of complete emptying after the bowel movement").
  Baseline was defined as the average number of CSBMs per day during the 2 weeks prior to receiving study drug (Day 1 to Day 15).
Time Frame: Baseline and 24 hours post-dose
Population: Intent-to-treat population; LOCF imputation was used
Measure: Mean (Standard Deviation); unit: complete spontaneous bowel movements/day
Arm/Group | Pooled Placebo | Naldemedine 0.01 mg | Naldemedine 0.03 mg | Naldemedine 0.1 mg | Naldemedine 0.3 mg | Naldemedine 1 mg | Naldemedine 3 mg
Number analyzed (Participants) | 18 | 9 | 9 | 9 | 9 | 9 | 9
complete spontaneous bowel movements/day
  Baseline | 0.03 (0.06) | 0.07 (0.09) | 0.07 (0.08) | 0.06 (0.10) | 0.01 (0.03) | 0.03 (0.04) | 0.10 (0.07)
  24 hours post-dose | 0.06 (0.24) | 0.00 (0.00) | 0.11 (0.33) | 0.22 (0.44) | 0.11 (0.33) | 2.44 (2.55) | 3.00 (3.20)
  Change from Baseline to 24 hours post-dose | 0.02 (0.25) | -0.07 (0.09) | 0.04 (0.29) | 0.16 (0.44) | 0.10 (0.34) | 2.42 (2.55) | 2.90 (3.24)
Statistical Analysis 1: Comparison: Pooled Placebo vs Naldemedine 0.01 mg; Test type: Superiority or Other; p = 0.6269, ANCOVA; P-values are from a non-parametric rank ANCOVA model with effects for dose group and gender, and baseline number of CSBMs as a covariate
Statistical Analysis 2: Comparison: Pooled Placebo vs Naldemedine 0.03 mg; Test type: Superiority or Other; p = 0.7456, ANCOVA; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Pooled Placebo vs Naldemedine 0.1 mg; Test type: Superiority or Other; p = 0.1968, ANCOVA; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Pooled Placebo vs Naldemedine 0.3 mg; Test type: Superiority or Other; p = 0.8708, ANCOVA; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: Pooled Placebo vs Naldemedine 1 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 6: Comparison: Pooled Placebo vs Naldemedine 3 mg; Test type: Superiority or Other; p = 0.0002, ANCOVA; [statistical method as in outcome 6, analysis 1]

7. Secondary Outcome: Change From Baseline to 48 Hours Post-dose in Number of Complete Spontaneous Bowel Movements (CSBMs) Per Day
Description: Participants completed a bowel function assessment daily diary to record information about bowel movements and constipation. A complete spontaneous bowel movement was defined as a bowel movement where no laxative or enema was used and the bowel movement resulted in a sensation of complete evacuation (based on the question of "having a feeling of complete emptying after the bowel movement").
  Baseline was defined as the average number of CSBMs per day during the 2 weeks prior to receiving study drug (Day 1 to Day 15). Forty-eight hours post-dose was defined as the average number of CSBMs per day from 0 to 48 hours post-dose.
Time Frame: Baseline and 48 hours post-dose
Population: Intent-to-treat population; LOCF imputation was used
Measure: Mean (Standard Deviation); unit: complete spontaneous bowel movements/day
Arm/Group | Pooled Placebo | Naldemedine 0.01 mg | Naldemedine 0.03 mg | Naldemedine 0.1 mg | Naldemedine 0.3 mg | Naldemedine 1 mg | Naldemedine 3 mg
Number analyzed (Participants) | 18 | 9 | 9 | 9 | 9 | 9 | 9
complete spontaneous bowel movements/day
  Baseline | 0.03 (0.06) | 0.07 (0.09) | 0.07 (0.08) | 0.06 (0.10) | 0.01 (0.03) | 0.03 (0.04) | 0.10 (0.07)
  48 hours post-dose | 0.08 (0.19) | 0.17 (0.25) | 0.17 (0.25) | 0.17 (0.35) | 0.06 (0.17) | 1.39 (1.34) | 1.61 (1.52)
  Change from baseline to 48 hours post-dose | 0.05 (0.16) | 0.10 (0.18) | 0.10 (0.25) | 0.10 (0.34) | 0.04 (0.17) | 1.36 (1.34) | 1.51 (1.56)
Statistical Analysis 1: Comparison: Pooled Placebo vs Naldemedine 0.01 mg; Test type: Superiority or Other; p = 0.6131, ANCOVA; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Pooled Placebo vs Naldemedine 0.03 mg; Test type: Superiority or Other; p = 0.9293, ANCOVA; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Pooled Placebo vs Naldemedine 0.1 mg; Test type: Superiority or Other; p = 0.7990, ANCOVA; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Pooled Placebo vs Naldemedine 0.3 mg; Test type: Superiority or Other; p = 0.7674, ANCOVA; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: Pooled Placebo vs Naldemedine 1 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 6: Comparison: Pooled Placebo vs Naldemedine 3 mg; Test type: Superiority or Other; p = 0.0018, ANCOVA; [statistical method as in outcome 6, analysis 1]

8. Secondary Outcome: Time to First Spontaneous Bowel Movement
Description: The time to first SBM during the Study Drug Administration Period was summarized using Kaplan-Meier estimates. Each participant's first SBM was counted as an event and the time to first SBM after dosing was calculated from the date and time of first dosing until the date and time of first SBM. Participants who dropped out or were lost to follow-up before the first SBM were censored.
Time Frame: From first dose on Day 15 through Day 17
Population: Intent-to-treat population
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Pooled Placebo | Naldemedine 0.01 mg | Naldemedine 0.03 mg | Naldemedine 0.1 mg | Naldemedine 0.3 mg | Naldemedine 1 mg | Naldemedine 3 mg
Number analyzed (Participants) | 18 | 9 | 9 | 9 | 9 | 9 | 9
hours | 27.2 [12.4 to NA] — Could not be estimated due to the low number of events | 37.0 [25.8 to NA] — Could not be estimated due to the low number of events | 13.9 [8.2 to NA] — Could not be estimated due to the low number of events | NA [3.3 to NA] — Could not be estimated due to the low number of events | 4.7 [2.8 to 6.2] | 1.4 [1.0 to 2.3] | 0.7 [0.6 to 0.8]
Statistical Analysis 1: Comparison: Pooled Placebo vs Naldemedine 0.01 mg; Test type: Superiority or Other; p = 0.7434, Log Rank; P-values were obtained from the log-rank test stratified by Gender; Hazard Ratio (HR) = 1.29, 95% CI 2-sided [0.42 to 3.92]
Statistical Analysis 2: Comparison: Pooled Placebo vs Naldemedine 0.03 mg; Test type: Superiority or Other; p = 0.4449, Log Rank; P-values were obtained from the log-rank test stratified by Gender; Hazard Ratio (HR) = 1.54, 95% CI 2-sided [0.54 to 4.42]
Statistical Analysis 3: Comparison: Pooled Placebo vs Naldemedine 0.1 mg; Test type: Superiority or Other; p = 0.8129, Log Rank; P-values were obtained from the log-rank test stratified by Gender; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.27 to 2.72]
Statistical Analysis 4: Comparison: Pooled Placebo vs Naldemedine 0.3 mg; Test type: Superiority or Other; p = 0.0005, Log Rank; P-values were obtained from the log-rank test stratified by Gender; Hazard Ratio (HR) = 7.52, 95% CI 2-sided [2.29 to 24.72]
Statistical Analysis 5: Comparison: Pooled Placebo vs Naldemedine 1 mg; Test type: Superiority or Other; p < 0.0001, Log Rank; P-values were obtained from the log-rank test stratified by Gender; Hazard Ratio (HR) = 9.93, 95% CI 2-sided [3.09 to 31.89]
Statistical Analysis 6: Comparison: Pooled Placebo vs Naldemedine 3 mg; Test type: Superiority or Other; p < 0.0001, Log Rank; P-values were obtained from the log-rank test stratified by Gender; Hazard Ratio (HR) = 202272814. — Hazard Ratio is infinite due to small range of observed times in 3 mg group that has no overlap with the Placebo group

9. Secondary Outcome: Time to First Bowel Movement
Description: The time to first BM during the Study Drug Administration Period was summarized using Kaplan-Meier estimates. Each participant's first BM was counted as an event and the time to first BM after dosing was calculated from the date and time of first dosing until the date and time of first BM. Participants who dropped out or were lost to follow-up before the first BM were censored.
Time Frame: From first dose on Day 15 through Day 17
Population: Intent-to-treat population
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Pooled Placebo | Naldemedine 0.01 mg | Naldemedine 0.03 mg | Naldemedine 0.1 mg | Naldemedine 0.3 mg | Naldemedine 1 mg | Naldemedine 3 mg
Number analyzed (Participants) | 18 | 9 | 9 | 9 | 9 | 9 | 9
hours | 27.2 [12.4 to NA] — Could not be estimated due to the low number of events | 28.4 [25.8 to 43.0] | 13.9 [8.2 to NA] — Could not be estimated due to the low number of events | 25.1 [3.3 to 57.3] | 4.7 [2.8 to 6.2] | 1.4 [1.0 to 2.3] | 0.7 [0.6 to 0.8]
Statistical Analysis 1: Comparison: Pooled Placebo vs Naldemedine 0.01 mg; Test type: Superiority or Other; p = 0.4923, Log Rank; P-values are from the log rank test stratified by gender; Hazard Ratio (HR) = 1.51, 95% CI 2-sided [0.53 to 4.28]
Statistical Analysis 2: Comparison: Pooled Placebo vs Naldemedine 0.03 mg; Test type: Superiority or Other; p = 0.5479, Log Rank; P-values are from the log rank test stratified by gender; Hazard Ratio (HR) = 1.45, 95% CI 2-sided [0.52 to 4.06]
Statistical Analysis 3: Comparison: Pooled Placebo vs Naldemedine 0.1 mg; Test type: Superiority or Other; p = 0.5060, Log Rank; P-values are from the log rank test stratified by gender; Hazard Ratio (HR) = 1.44, 95% CI 2-sided [0.56 to 3.67]
Statistical Analysis 4: Comparison: Pooled Placebo vs Naldemedine 0.3 mg; Test type: Superiority or Other; p = 0.0005, Log Rank; P-values are from the log rank test stratified by gender; Hazard Ratio (HR) = 7.36, 95% CI 2-sided [2.27 to 23.90]
Statistical Analysis 5: Comparison: Pooled Placebo vs Naldemedine 1 mg; Test type: Superiority or Other; p < 0.0001, Log Rank; P-values are from the log rank test stratified by gender; Hazard Ratio (HR) = 9.54, 95% CI 2-sided [3.00 to 30.35]
Statistical Analysis 6: Comparison: Pooled Placebo vs Naldemedine 3 mg; Test type: Superiority or Other; p < 0.0001, Log Rank; P-values are from the log rank test stratified by gender; Hazard Ratio (HR) = 192233779 — Hazard Ratio is infinite due to small range of observed times in 3 mg group that has no overlap with the Placebo group

10. Secondary Outcome: Time to First Complete Spontaneous Bowel Movement
Description: The time to first CSBM during the Study Drug Administration Period was summarized using Kaplan-Meier estimates. Each participant's first CSBM was counted as an event and the time to first CSBM after dosing was calculated from the date and time of first dosing until the date and time of first CSBM. Participants who dropped out or were lost to follow-up before the first CSBM were censored.
Time Frame: From first dose on Day 15 through Day 17
Population: Intent-to-treat population
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Pooled Placebo | Naldemedine 0.01 mg | Naldemedine 0.03 mg | Naldemedine 0.1 mg | Naldemedine 0.3 mg | Naldemedine 1 mg | Naldemedine 3 mg
Number analyzed (Participants) | 18 | 9 | 9 | 9 | 9 | 9 | 9
hours | NA [NA to NA] — Could not be estimated due to the low number of events | NA [37.0 to NA] — Could not be estimated due to the low number of events | NA [37.7 to NA] — Could not be estimated due to the low number of events | NA [NA to NA] — Could not be estimated due to the low number of events | NA [NA to NA] — Could not be estimated due to the low number of events | 1.7 [1.3 to 2.3] | 0.8 [0.6 to 25.8]
Statistical Analysis 1: Comparison: Pooled Placebo vs Naldemedine 0.01 mg; Test type: Superiority or Other; p = 0.1523, Log Rank; P-values are from the log rank test stratified by gender; Hazard Ratio (HR) = 3.45, 95% CI 2-sided [0.62 to 19.35]
Statistical Analysis 2: Comparison: Pooled Placebo vs Naldemedine 0.03 mg; Test type: Superiority or Other; p = 0.0856, Log Rank; P-values are from the log rank test stratified by gender; Hazard Ratio (HR) = 4.55, 95% CI 2-sided [0.76 to 27.07]
Statistical Analysis 3: Comparison: Pooled Placebo vs Naldemedine 0.1 mg; Test type: Superiority or Other; p = 0.5284, Log Rank; P-values are from the log rank test stratified by gender; Hazard Ratio (HR) = 1.81, 95% CI 2-sided [0.30 to 10.98]
Statistical Analysis 4: Comparison: Pooled Placebo vs Naldemedine 0.3 mg; Test type: Superiority or Other; p = 0.8594, Log Rank; P-values are from the log rank test stratified by gender; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.09 to 8.66]
Statistical Analysis 5: Comparison: Pooled Placebo vs Naldemedine 1 mg; Test type: Superiority or Other; p < 0.0001, Log Rank; P-values are from the log rank test stratified by gender; Hazard Ratio (HR) = 59.34, 95% CI 2-sided [6.55 to 537.38]
Statistical Analysis 6: Comparison: Pooled Placebo vs Naldemedine 3 mg; Test type: Superiority or Other; p = 0.0007, Log Rank; P-values are from the log rank test stratified by gender; Hazard Ratio (HR) = 10.99, 95% CI 2-sided [2.30 to 52.57]

11. Secondary Outcome: Change From Baseline in Straining During Bowel Movements
Description: Straining during BMs was graded using the following scale: 0 = Absent; 1 = Mild; 2 = Moderate; 3 = Severe; 4 = Very Severe.
  Baseline was defined as the average straining score of all BMs prior to receiving study drug (Day 1 to Day 15). The straining score at 24 and 48 hours post-dose was calculated as the average straining score from all bowel movements from 0 to 24 and 0 to 48 hours post-dose, respectively.
Time Frame: Baseline, 24 hours post-dose and 48 hours post-dose
Population: Intent-to-treat population with available data at each time point
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pooled Placebo | Naldemedine 0.01 mg | Naldemedine 0.03 mg | Naldemedine 0.1 mg | Naldemedine 0.3 mg | Naldemedine 1 mg | Naldemedine 3 mg
Number analyzed (Participants) | 18 | 9 | 9 | 9 | 9 | 9 | 9
units on a scale
  Baseline | 2.2 (0.71) | 2.0 (0.78) | 2.2 (0.68) | 1.9 (0.90) | 2.0 (1.08) | 2.5 (0.97) | 1.7 (0.99)
  Change from Baseline to 24 hours post-dose: number analyzed (Participants) | 8 | 1 | 5 | 4 | 8 | 9 | 9
  Change from Baseline to 24 hours post-dose | 0.8 (0.76) | -0.8 (NA) — Standard deviation cannot be calculated when n=1 | -0.2 (0.88) | -0.7 (0.43) | -0.1 (0.89) | -0.5 (1.37) | -0.9 (1.64)
  Change from Baseline to 48 hours post-dose: number analyzed (Participants) | 6 | 7 | 4 | 4 | 1 | 3 | 3
  Change from Baseline to 48 hours post-dose | 0.5 (0.87) | 0.2 (0.74) | 0.4 (0.80) | -0.6 (0.67) | 0.1 (NA) — Standard deviation cannot be calculated when n=1 | -0.4 (0.42) | -1.4 (1.40)

12. Secondary Outcome: Change From Baseline to 24 Hours Post-dose in Number of Complete Bowel Movements Per Day
Description: A complete bowel movement (CBM) was defined as a bowel movement that resulted in a sensation of complete evacuation based on the question "Did you have a feeling of complete emptying after the bowel movement?" Baseline was defined as the average number of CBMs per day prior to receiving study drug (Day 1 to Day 15).
Time Frame: Baseline and 24 hours post-dose
Population: Intent-to-treat population; LOCF imputation was used
Measure: Mean (Standard Deviation); unit: complete bowel movements / day
Arm/Group | Pooled Placebo | Naldemedine 0.01 mg | Naldemedine 0.03 mg | Naldemedine 0.1 mg | Naldemedine 0.3 mg | Naldemedine 1 mg | Naldemedine 3 mg
Number analyzed (Participants) | 18 | 9 | 9 | 9 | 9 | 9 | 9
complete bowel movements / day
  Baseline | 0.13 (0.16) | 0.13 (0.14) | 0.11 (0.09) | 0.14 (0.12) | 0.04 (0.06) | 0.12 (0.15) | 0.19 (0.15)
  24 hours post-dose | 0.06 (0.24) | 0.00 (0.00) | 0.11 (0.33) | 0.22 (0.44) | 0.11 (0.33) | 2.44 (2.55) | 3.00 (3.20)
  Change from baseline to 24 hours post-dose | -0.07 (0.20) | -0.13 (0.14) | 0.01 (0.31) | 0.09 (0.45) | 0.07 (0.35) | 2.32 (2.61) | 2.81 (3.21)
Statistical Analysis 1: Comparison: Pooled Placebo vs Naldemedine 0.01 mg; Test type: Superiority or Other; p = 0.5054, ANCOVA; P-values were obtained from a non-parametric rank ANCOVA model with effects for dose group and gender, and baseline number of CBMs as a covariate
Statistical Analysis 2: Comparison: Pooled Placebo vs Naldemedine 0.03 mg; Test type: Superiority or Other; p = 0.9688, ANCOVA; [statistical method as in outcome 12, analysis 1]
Statistical Analysis 3: Comparison: Pooled Placebo vs Naldemedine 0.1 mg; Test type: Superiority or Other; p = 0.6963, ANCOVA; [statistical method as in outcome 12, analysis 1]
Statistical Analysis 4: Comparison: Pooled Placebo vs Naldemedine 0.3 mg; Test type: Superiority or Other; p = 0.9599, ANCOVA; [statistical method as in outcome 12, analysis 1]
Statistical Analysis 5: Comparison: Pooled Placebo vs Naldemedine 1 mg; Test type: Superiority or Other; p = 0.0001, ANCOVA; [statistical method as in outcome 12, analysis 1]
Statistical Analysis 6: Comparison: Pooled Placebo vs Naldemedine 3 mg; Test type: Superiority or Other; p = 0.0006, ANCOVA; [statistical method as in outcome 12, analysis 1]

13. Secondary Outcome: Change From Baseline to 48 Hours Post-dose in Number of Complete Bowel Movements Per Day
Description: A complete bowel movement (CBM) was defined as a bowel movement that resulted in a sensation of complete evacuation based on the question "Did you have a feeling of complete emptying after the bowel movement?" Baseline was defined as the average number of CBMs per day prior to receiving study drug (Day 1 to 15). Forty-eight hours post-dose was calculated as the average number of CBMs per day from 0 to 48 hours post-dose.
Time Frame: Baseline and 48 hours post-dose
Population: Intent-to-treat population; LOCF imputation was used
Measure: Mean (Standard Deviation); unit: complete bowel movements / day
Arm/Group | Pooled Placebo | Naldemedine 0.01 mg | Naldemedine 0.03 mg | Naldemedine 0.1 mg | Naldemedine 0.3 mg | Naldemedine 1 mg | Naldemedine 3 mg
Number analyzed (Participants) | 18 | 9 | 9 | 9 | 9 | 9 | 9
complete bowel movements / day
  Baseline | 0.13 (0.16) | 0.13 (0.14) | 0.11 (0.09) | 0.14 (0.12) | 0.04 (0.06) | 0.12 (0.15) | 0.19 (0.15)
  48 hours post-dose | 0.08 (0.19) | 0.17 (0.25) | 0.17 (0.25) | 0.22 (0.36) | 0.06 (0.17) | 1.39 (1.34) | 1.61 (1.52)
  Change from Baseline to 48 hours post-dose | -0.04 (0.17) | 0.04 (0.15) | 0.06 (0.28) | 0.09 (0.38) | 0.01 (0.19) | 1.27 (1.38) | 1.42 (1.53)
Statistical Analysis 1: Comparison: Pooled Placebo vs Naldemedine 0.01 mg; Test type: Superiority or Other; p = 0.3441, ANCOVA; [statistical method as in outcome 12, analysis 1]
Statistical Analysis 2: Comparison: Pooled Placebo vs Naldemedine 0.03 mg; Test type: Superiority or Other; p = 0.7159, ANCOVA — P-values were obtained from a non-parametric rank ANCOVA model with effects for dose group and gender, and baseline number of CBMs as a covariate
Statistical Analysis 3: Comparison: Pooled Placebo vs Naldemedine 0.1 mg; Test type: Superiority or Other; p = 0.7342, ANCOVA; [statistical method as in outcome 12, analysis 1]
Statistical Analysis 4: Comparison: Pooled Placebo vs Naldemedine 0.3 mg; Test type: Superiority or Other; p = 0.8714, ANCOVA; [statistical method as in outcome 12, analysis 1]
Statistical Analysis 5: Comparison: Pooled Placebo vs Naldemedine 1 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 12, analysis 1]
Statistical Analysis 6: Comparison: Pooled Placebo vs Naldemedine 3 mg; Test type: Superiority or Other; p = 0.0006, ANCOVA; [statistical method as in outcome 12, analysis 1]

14. Secondary Outcome: Change From Baseline in Abdominal Bloating
Description: Participants were asked to rate their abdominal bloating for the past 24 hours using the following scale:
  0 = Absent; 1 = Mild; 2 = Moderate; 3 = Severe; 4 = Very Severe. Baseline was defined as the average abdominal bloating score prior to receiving study drug (Day 1 to Day 15). Abdominal bloating at 24 hours and 48 hours post-dose was calculated as the mean score from 0 to 24 and 0 to 48 hours post-dose respectively.
Time Frame: Baseline, 24 hours post-dose and 48 hours post-dose
Population: Intent-to-treat population with available data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pooled Placebo | Naldemedine 0.01 mg | Naldemedine 0.03 mg | Naldemedine 0.1 mg | Naldemedine 0.3 mg | Naldemedine 1 mg | Naldemedine 3 mg
Number analyzed (Participants) | 18 | 9 | 9 | 9 | 9 | 9 | 9
units on a scale
  Baseline | 2.0 (0.65) | 1.4 (0.95) | 1.5 (0.69) | 1.7 (0.87) | 1.7 (0.66) | 2.5 (0.64) | 1.3 (0.65)
  Change from Baseline to 24 hours post-dose: number analyzed (Participants) | 8 | 1 | 5 | 4 | 8 | 9 | 9
  Change from Baseline to 24 hours post-dose | 0.0 (0.83) | 0.0 (NA) — Cannot be calculated when n=1 | 0.2 (1.09) | -0.2 (1.03) | 0.3 (0.69) | -0.5 (0.91) | 0.7 (1.53)
  Change from Baseline to 48 hours post-dose: number analyzed (Participants) | 6 | 7 | 4 | 4 | 1 | 3 | 3
  Change from Baseline to 48 hours post-dose | -0.5 (0.54) | 0.1 (0.86) | 0.2 (1.17) | 0.1 (0.89) | 0.4 (NA) — Cannot be calculated when n=1 | -0.8 (0.5) | -0.2 (1.95)

15. Secondary Outcome: Change From Baseline in Abdominal Discomfort
Description: Participants were asked to rate their abdominal discomfort for the past 24 hours using the following scale:
  0 = Absent; 1 = Mild; 2 = Moderate; 3 = Severe; 4 = Very Severe. Baseline was defined as the average abdominal discomfort score prior to receiving study drug (Day 1 to Day 15). Abdominal discomfort at 24 hours and 48 hours post-dose was calculated as the mean score from 0 to 24 and 0 to 48 hours post-dose respectively.
Time Frame: Baseline, 24 hours post-dose and 48 hours post-dose
Population: Intent-to-treat population with available data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pooled Placebo | Naldemedine 0.01 mg | Naldemedine 0.03 mg | Naldemedine 0.1 mg | Naldemedine 0.3 mg | Naldemedine 1 mg | Naldemedine 3 mg
Number analyzed (Participants) | 18 | 9 | 9 | 9 | 9 | 9 | 9
units on a scale
  Baseline | 2.1 (0.63) | 1.5 (0.98) | 2.0 (0.75) | 2.0 (0.74) | 1.9 (0.81) | 2.6 (0.77) | 1.7 (0.77)
  Change from Baseline to 24 hours post-dose: number analyzed (Participants) | 8 | 1 | 5 | 4 | 8 | 9 | 9
  Change from Baseline to 24 hours post-dose | -0.2 (0.78) | -0.8 (NA) — Cannot be calculated when n=1 | -0.5 (0.80) | -0.7 (1.30) | 0.3 (0.60) | -0.1 (0.96) | 1.3 (0.90)
  Change from Baseline to 48 hours post-dose: number analyzed (Participants) | 6 | 7 | 4 | 4 | 1 | 3 | 3
  Change from Baseline to 48 hours post-dose | -0.4 (0.67) | -0.3 (1.00) | -0.2 (1.00) | -0.4 (0.44) | 1.1 (NA) — Cannot be calculated when n=1 | -1.1 (1.07) | -0.1 (1.59)

16. Secondary Outcome: Change From Baseline in BM Consistency
Description: Consistency of BMs was measured using the Bristol Stool Scale, as follows:
  1 = separate hard lumps like nuts; 2 = sausage shaped but lumpy; 3 = like a sausage, but with cracks on its surface; 4 = like a sausage or a snake, smooth and soft; 5 = soft blobs and with clear-cut edges; 6 = floppy pieces with ragged edges/mushy stool; 7 = watery, no solid pieces, entirely liquid.
  Baseline was defined as the average consistency of BMs prior to receiving study drug (Day 1 to Day 15). BM consistency at 24 hours and 48 hours post-dose was calculated as the average scores from all bowel movements from 0 to 24 and 0 to 48 hours post-dose, respectively.
Time Frame: Baseline, 24 hours post-dose and 48 hours post-dose
Population: Intent-to-treat population with available data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pooled Placebo | Naldemedine 0.01 mg | Naldemedine 0.03 mg | Naldemedine 0.1 mg | Naldemedine 0.3 mg | Naldemedine 1 mg | Naldemedine 3 mg
Number analyzed (Participants) | 18 | 9 | 9 | 9 | 9 | 9 | 9
units on a scale
  Baseline | 2.9 (1.24) | 3.2 (1.13) | 2.2 (1.12) | 3.0 (1.71) | 3.2 (1.33) | 3.2 (2.06) | 2.2 (0.81)
  Change from Baseline to 24 hours post-dose: number analyzed (Participants) | 8 | 1 | 5 | 4 | 8 | 9 | 9
  Change from Baseline to 24 hours post-dose | -1.4 (1.09) | -3.0 (NA) — Cannot be calculated when n=1 | -0.0 (0.24) | -1.4 (1.56) | 1.5 (1.44) | 1.9 (3.27) | 4.1 (1.07)
  Change from Baseline to 48 hours post-dose: number analyzed (Participants) | 6 | 7 | 4 | 4 | 1 | 3 | 3
  Change from Baseline to 48 hours post-dose | -1.0 (1.45) | 0.2 (2.45) | -0.3 (1.43) | -1.0 (2.00) | 0.6 (NA) — Cannot be calculated when n=1 | 0.7 (3.66) | 2.5 (1.88)

17. Secondary Outcome: Change From Baseline in Number of False Start Bowel Movements Per Day
Description: A false start was defined as any attempted, but unsuccessful bowel movement (no solid or liquid fecal material was excreted) based on the question "In the past 24 hours, how many times did you try to have a bowel movement but were unsuccessful?" Baseline was defined as the average number of false start BMs per day prior to receiving study drug (Day 1 to Day 15).
  The number of false start BMs per day at 24 hours and 48 hours post-dose was calculated as is the average number of false start BMs per day from 0 to 24 and 0 to 48 hours post-dose, respectively.
Time Frame: Baseline, 24 hours post-dose and 48 hours post-dose
Population: Intent-to-treat population; LOCF imputation was used
Measure: Mean (Standard Deviation); unit: false start bowel movements / day
Arm/Group | Pooled Placebo | Naldemedine 0.01 mg | Naldemedine 0.03 mg | Naldemedine 0.1 mg | Naldemedine 0.3 mg | Naldemedine 1 mg | Naldemedine 3 mg
Number analyzed (Participants) | 18 | 9 | 9 | 9 | 9 | 9 | 9
false start bowel movements / day
  Baseline | 0.56 (0.86) | 0.67 (1.00) | 0.67 (1.12) | 0.22 (0.44) | 0.56 (1.01) | 0.00 (0.00) | 0.33 (0.50)
  Change from Baseline to 24 hours post-dose | 0.28 (0.89) | 0.44 (1.33) | -0.11 (1.17) | 0.00 (0.50) | -0.11 (0.60) | 2.56 (3.81) | 0.78 (1.79)
  Change from Baseline to 48 hours post-dose | 0.25 (0.69) | 0.28 (1.18) | 0.22 (1.48) | 0.00 (0.50) | -0.06 (0.58) | 1.61 (2.42) | 0.44 (0.77)

18. Secondary Outcome: Change From Baseline in the Number of Bowel Movements With No Straining Per Day
Description: Straining during BMs was graded using the following scale:
  0 = Absent; 1 = Mild; 2 = Moderate; 3 = Severe; 4 = Very Severe. A BM without straining was defined as a BM with a straining score = 0.
  Baseline was defined as the average number of BMs without straining per day prior to receiving study drug (Day 1 to Day 15). The number of BMs without straining per day at 24 hours and 48 hours post-dose was calculated as the average number of BMs with no straining per day from 0 to 24 hours and 0 to 48 hours post-dose, respectively.
Time Frame: Baseline, 24 hours post-dose and 48 hours post-dose
Population: Intent-to-treat population; LOCF imputation was used
Measure: Mean (Standard Deviation); unit: bowel movements with no straining / day
Arm/Group | Pooled Placebo | Naldemedine 0.01 mg | Naldemedine 0.03 mg | Naldemedine 0.1 mg | Naldemedine 0.3 mg | Naldemedine 1 mg | Naldemedine 3 mg
Number analyzed (Participants) | 18 | 9 | 9 | 9 | 9 | 9 | 9
bowel movements with no straining / day
  Baseline | 0.03 (0.07) | 0.09 (0.11) | 0.05 (0.09) | 0.03 (0.07) | 0.05 (0.07) | 0.03 (0.05) | 0.07 (0.11)
  Change from Baseline to 24 hours post-dose | -0.03 (0.07) | -0.09 (0.11) | 0.06 (0.36) | -0.03 (0.07) | 0.28 (0.71) | 0.41 (0.74) | 3.37 (2.16)
  Change from Baseline to 48 hours post-dose | -0.01 (0.14) | -0.03 (0.13) | 0.01 (0.21) | -0.03 (0.07) | 0.12 (0.36) | 0.19 (0.38) | 1.76 (1.02)

19. Secondary Outcome: Change From Baseline in Number of Rescue Medications Used Per Day
Description: Baseline was defined as the average number of rescue medications used per day prior to receiving study drug (Day 1 to Day 15). The number of rescue medications used per day at 24 hours and 48 hours post-dose was calculated as the average number of rescue medications used per day from 0 to 24 hours and 0 to 48 hours post-dose, respectively.
Time Frame: Baseline, 24 hours post-dose and 48 hours post-dose
Population: Intent-to-treat population; LOCF imputation was used
Measure: Mean (Standard Deviation); unit: rescue medications / day
Arm/Group | Pooled Placebo | Naldemedine 0.01 mg | Naldemedine 0.03 mg | Naldemedine 0.1 mg | Naldemedine 0.3 mg | Naldemedine 1 mg | Naldemedine 3 mg
Number analyzed (Participants) | 18 | 9 | 9 | 9 | 9 | 9 | 9
rescue medications / day
  Baseline | 0.31 (0.36) | 0.18 (0.21) | 0.36 (0.43) | 0.53 (0.68) | 0.52 (0.84) | 0.28 (0.36) | 0.20 (0.24)
  Change from Baseline to 24 hours post-dose | -0.04 (0.70) | -0.18 (0.21) | -0.36 (0.43) | 0.02 (1.13) | -0.52 (0.84) | -0.28 (0.36) | -0.20 (0.24)
  Change from Baseline to 48 hours post-dose | -0.04 (0.51) | -0.01 (0.36) | -0.25 (0.37) | 0.08 (0.80) | -0.52 (0.84) | -0.23 (0.38) | -0.20 (0.24)

20. Secondary Outcome: Percentage of Participants With Clinical Opiate Withdrawal Scale (COWS) Score > 8 at Any Time During the Study
Description: The COWS assessment consisted of 11 questions which rated the severity of opiate withdrawal symptoms, including resting pulse rate, gastrointestinal upset, sweating, restlessness, pupil size, tremor, anxiety or irritability, bone or joint aches, gooseflesh skin, yawning, and runny nose or tearing. Each symptom was rated on a scale from 0 (not present) to 4 or 5 (most severe). The total score was calculated by summing the 11 individual scores and ranged from 0 (no withdrawal symptoms) to 48 (worst symptoms).
Time Frame: The COWS assessments were performed at Screening, on Day 14, Day 15 (pre-dose and 1, 2, 3, 4, 5, 6 and 8 hours post-dose, and at unscheduled times as signs or symptoms indicate), on Days 16 and 17, and on Day 24/End of Study.
Population: Safety population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pooled Placebo | Naldemedine 0.01 mg | Naldemedine 0.03 mg | Naldemedine 0.1 mg | Naldemedine 0.3 mg | Naldemedine 1 mg | Naldemedine 3 mg
Number analyzed (Participants) | 18 | 9 | 9 | 9 | 9 | 9 | 9
percentage of participants | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 33.6] | 11.1 [0.3 to 48.2] | 66.7 [29.9 to 92.5]

21. Secondary Outcome: Percentage of Participants With Webster Opiate Withdrawal Scale (WOWS) Score > 8 at Any Time During the Study
Description: The Webster Opiate Withdrawal Scale (WOWS) assessment consisted of 7 questions which rate the severity of opiate withdrawal symptoms, including sweating, sleep, bone or joint aches, runny nose or tearing, gastrointestinal upset, anxiety or irritability and gooseflesh skin. Each symptom was rated on a scale from 0 (not present/no issues) to 4 or 5 (severe). The total score was calculated by summing the 7 individual scores and ranged from 0 (no withdrawal symptoms) to 29 (worst symptoms).
Time Frame: The WOWS assessment was performed at Screening, Day 14, Day 15 at pre-dose , and 24 and 48 hours post-dose and at the Follow-up/End of Study visit (Day 24).
Population: Safety population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pooled Placebo | Naldemedine 0.01 mg | Naldemedine 0.03 mg | Naldemedine 0.1 mg | Naldemedine 0.3 mg | Naldemedine 1 mg | Naldemedine 3 mg
Number analyzed (Participants) | 18 | 9 | 9 | 9 | 9 | 9 | 9
percentage of participants | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 33.6] | 11.1 [0.3 to 48.2] | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 33.6]

22. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Naldemedine and Metabolite Nor-S-297995
Description: The plasma concentration of naldemedine and its metabolite Nor-S-297995 were measured by liquid chromatography/tandem mass spectrometry (LC/MS/MS) method.
Time Frame: Blood samples were collected predose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, and 72 hours post-dose.
Population: The pharmacokinetic (PK) analysis population included all randomized participants who received study drug and had at least one post-dose PK assessment completed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Naldemedine 0.01 mg | Naldemedine 0.03 mg | Naldemedine 0.1 mg | Naldemedine 0.3 mg | Naldemedine 1 mg | Naldemedine 3 mg
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9
ng/mL
  Naldemedine | 0.0837 (29.6) | 0.290 (28.9) | 1.00 (28.4) | 3.12 (30.2) | 9.68 (31.3) | 30.9 (44.2)
  Nor-S-297995 | NA (NA) — Nor-S-297995 could not be quantified | NA (NA) — Nor-S-297995 could not be quantified | 0.0713 (31.8) | 0.134 (27.6) | 0.526 (49.4) | 1.50 (53.3)

23. Secondary Outcome: Time to Maximum Observed Plasma Concentration of Naldemedine and Metabolite Nor-S-297995
Description: as for outcome 22
Time Frame: as for outcome 22
Population: PK population
Measure: Median (Full Range); unit: hours
Arm/Group | Naldemedine 0.01 mg | Naldemedine 0.03 mg | Naldemedine 0.1 mg | Naldemedine 0.3 mg | Naldemedine 1 mg | Naldemedine 3 mg
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9
hours
  Naldemedine | 0.75 [0.5 to 3.0] | 1.0 [0.5 to 4.0] | 2.5 [0.5 to 5.0] | 1.0 [0.72 to 3.0] | 1.0 [0.75 to 2.0] | 0.75 [0.50 to 1.0]
  Nor-S-297995 | NA [NA to NA] — Nor-S-297995 could not be quantified | NA [NA to NA] — Nor-S-297995 could not be quantified | 5.0 [2.5 to 12] | 4.1 [3.0 to 8.0] | 8.0 [4.0 to 12] | 5.0 [3.0 to 10]

24. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Time of Last Measurable Concentration of Naldemedine and Metabolite Nor-S-297995
Description: The plasma concentration of naldemedine and its metabolite Nor-S-297995 were measured by liquid chromatography/tandem mass spectrometry (LC/MS/MS) method. Area under the plasma concentration versus time curve from time zero to the last sampling time at which concentrations were at or above the limit of quantitation, calculated using the linear trapezoidal rule for increasing concentrations and the logarithmic rule for decreasing concentrations (Linear Up/ Log Down).
Time Frame: as for outcome 22
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL)
Arm/Group | Naldemedine 0.01 mg | Naldemedine 0.03 mg | Naldemedine 0.1 mg | Naldemedine 0.3 mg | Naldemedine 1 mg | Naldemedine 3 mg
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9
ng*hr/mL)
  Naldemedine | 0.5863 (34.3) | 2.111 (31.4) | 11.71 (21.4) | 31.29 (30.5) | 93.60 (34.6) | 218.2 (37.6)
  Nor-S-297995 | NA (NA) — Nor-S-297995 could not be quantified | NA (NA) — Nor-S-297995 could not be quantified | 0.5856 (232.7) | 1.869 (68.3) | 14.97 (76.3) | 41.94 (63.3)

25. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity for Naldemedine and Metabolite Nor-S-297995
Description: The plasma concentration of naldemedine and its metabolite Nor-S-297995 were measured by liquid chromatography/tandem mass spectrometry (LC/MS/MS) method. Area under the plasma concentration versus time curve from time zero to infinity, calculated using the formula: AUC0-inf = AUC0-t + Ct/λZ where Ct was the last measurable concentration and λZ was the apparent terminal elimination rate constant.
Time Frame: as for outcome 22
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Naldemedine 0.01 mg | Naldemedine 0.03 mg | Naldemedine 0.1 mg | Naldemedine 0.3 mg | Naldemedine 1 mg | Naldemedine 3 mg
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9
ng*hr/mL
  Naldemedine | 0.8023 (33.8) | 2.294 (30.2) | 12.04 (21.7) | 31.87 (29.9) | 94.53 (34.8) | 219.9 (37.8)
  Nor-S-297995 | NA (NA) — Nor-S-297995 could not be quantified | NA (NA) — Nor-S-297995 could not be quantified | 3.046 (63.0) | 4.515 (58.8) | 17.10 (73.4) | 44.91 (63.6)

26. Secondary Outcome: Apparent Elimination Half-life of Naldemedine and Metabolite Nor-S-297995
Description: The plasma concentration of naldemedine and its metabolite Nor-S-297995 were measured by liquid chromatography/tandem mass spectrometry (LC/MS/MS) method. The apparent elimination half-life was calculated using the formula t1/2,z = (ln2)/λZ
Time Frame: as for outcome 22
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Naldemedine 0.01 mg | Naldemedine 0.03 mg | Naldemedine 0.1 mg | Naldemedine 0.3 mg | Naldemedine 1 mg | Naldemedine 3 mg
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9
hours
  Naldemedine | 8.13 (58.3) | 7.46 (38.5) | 12.6 (35.6) | 12.2 (34.6) | 10.8 (20.9) | 11.6 (20.8)
  Nor-S-297995 | NA (NA) — Nor-S-297995 could not be quantified | NA (NA) — Nor-S-297995 could not be quantified | 24.6 (52.7) | 25.7 (61.8) | 16.0 (24.8) | 17.0 (18.1)

ADVERSE EVENTS:
Time Frame: From first dose of study drug on Day 15 up to Day 24 (10 days).
Groups:
- Naldemedine 1 mg: Participants received a single dose of 1mg naldemedine tablets administered on Day 15 under fasted conditions.
Arm/Group | Pooled Placebo | Naldemedine 0.01 mg | Naldemedine 0.03 mg | Naldemedine 0.1 mg | Naldemedine 0.3 mg | Naldemedine 1 mg | Naldemedine 3 mg
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 9/18 | 6/9 | 6/9 | 5/9 | 9/9 | 9/9 | 9/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pooled Placebo (N=18) | Naldemedine 0.01 mg (N=9) | Naldemedine 0.03 mg (N=9) | Naldemedine 0.1 mg (N=9) | Naldemedine 0.3 mg (N=9) | Naldemedine 1 mg (N=9) | Naldemedine 3 mg (N=9)
Abdominal pain (Gastrointestinal disorders) | 3 | 2 | 1 | 1 | 6 | 6 | 9
Nausea (Gastrointestinal disorders) | 3 | 4 | 0 | 0 | 1 | 7 | 6
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 2 | 3 | 8
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 3 | 6
Flatulence (Gastrointestinal disorders) | 2 | 2 | 0 | 0 | 2 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 2 | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tongue discolouration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 6
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Drug withdrawal syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Venipuncture site thrombosis (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infusion site rash (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 4 | 6
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 2 | 0 | 0 | 0 | 2 | 3
Headache (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 3
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Oxygen saturation decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 4
Cardiac murmur (Investigations) | 2 | 0 | 0 | 0 | 0 | 0 | 1
Blood glucose decreased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Blood prolactin increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Heart rate irregular (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pallor (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can embargo results from a PI's center until the combined results from the completed study have been published in full or the sponsor confirms there will be no multicenter study publication. Results communications must be provided to the sponsor for review at least 60 days before submission for publication. By written request, the sponsor can extend the embargo up to an additional 60 days. The sponsor cannot require changes to scientific content and cannot further extend the embargo.